CLINICAL TRIAL: NCT01531348
Title: Feasibility and Safety of Adult Human Bone Marrow-Derived Mesenchymal Stem Cells by Intravitreal Injection in Patients With Retinitis Pigmentosa
Brief Title: Intravitreal Injection of MSCs in Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, La-ongsri Atchaneeyasakul, Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RP-001
Record Dates: First submitted 2012-02-06; First posted 2012-02-10 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; Bone marrow-derived mesenchymal stem cells; Intravitreal injection
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BM-MSC (Experimental): Bone marrow-derived mesenchymal stem cells 1 million cells in balanced salt solution 100 microlitres will be injected into the vitreous cavity.
  Interventions: Other: BM-MSC

INTERVENTIONS:
Other: BM-MSC — Bone marrow-derived mesenchymal stem cells 1 million cells in balanced salt solution 100 microlitres will be injected into the vitreous cavity.

SUMMARY:
The purpose of this study is to determine the feasibility and safety of adult human bone marrow-derived mesenchymal stem cells by intravitreal injection in patients with retinitis pigmentosa.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is an inherited disorder of the photoreceptor cells in the retina. Patients may lose vision since they were young or later in life. Currently, there are more than 60 genes identified as the cause of this condition, one of which, RPE65, has been studied in several gene therapy trials for Leber congenital amaurosis with promising results. Another treatment approach for RP is stem cell therapy. Studies in animal models of RP have shown that subretinal injection of bone marrow-derived mesenchymal stem cells may delay degenerative changes of photoreceptor cells.

ELIGIBILITY:
Inclusion Criteria:

* Retinitis pigmentosa patients diagnosed by ophthalmologists
* Age 18-65 years old
* Central visual field less than or equal to 20 degrees
* Best corrected visual acuity less than 6/120 by Snellen visual acuity chart
* Electroretinogram nonrecordable or the amplitudes were less than 25% of normal

Exclusion Criteria:

* Other eye conditions that could mask the interpretation of the results
* Unable to return for follow up
* Underlying diseases including asthma, heart failure, myocardial infarction, liver failure, renal failure
* Pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in laser flare and cell measurements | up to 12 months

SECONDARY OUTCOMES:
Change from baseline in visual function tests | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: La-ongsri Atchaneeyasakul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Hartong DT, Berson EL, Dryja TP. Retinitis pigmentosa. Lancet. 2006 Nov 18;368(9549):1795-809. doi: 10.1016/S0140-6736(06)69740-7. PMID 17113430
- [Background] Kociok N. Can the injection of the patient's own bone marrow-derived stem cells preserve cone vision in retinitis pigmentosa and other diseases of the eye? Graefes Arch Clin Exp Ophthalmol. 2005 Mar;243(3):187-8. doi: 10.1007/s00417-004-1062-0. Epub 2004 Nov 23. No abstract available. PMID 15565292
- [Result] Arnhold S, Absenger Y, Klein H, Addicks K, Schraermeyer U. Transplantation of bone marrow-derived mesenchymal stem cells rescue photoreceptor cells in the dystrophic retina of the rhodopsin knockout mouse. Graefes Arch Clin Exp Ophthalmol. 2007 Mar;245(3):414-22. doi: 10.1007/s00417-006-0382-7. Epub 2006 Aug 4. PMID 16896916
- [Result] Wang S, Lu B, Girman S, Duan J, McFarland T, Zhang QS, Grompe M, Adamus G, Appukuttan B, Lund R. Non-invasive stem cell therapy in a rat model for retinal degeneration and vascular pathology. PLoS One. 2010 Feb 15;5(2):e9200. doi: 10.1371/journal.pone.0009200. PMID 20169166
- [Derived] Tuekprakhon A, Sangkitporn S, Trinavarat A, Pawestri AR, Vamvanij V, Ruangchainikom M, Luksanapruksa P, Pongpaksupasin P, Khorchai A, Dambua A, Boonchu P, Yodtup C, Uiprasertkul M, Sangkitporn S, Atchaneeyasakul LO. Intravitreal autologous mesenchymal stem cell transplantation: a non-randomized phase I clinical trial in patients with retinitis pigmentosa. Stem Cell Res Ther. 2021 Jan 9;12(1):52. doi: 10.1186/s13287-020-02122-7. PMID 33422139